CLINICAL TRIAL: NCT07098767
Title: Investigating the Reliability of Using Ultrasonography to Assess Swallowing Function in Patients With Dysphagia
Brief Title: SURE Trial: Swallowing Ultrasound Reliability Evaluation Trial
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202406013RINA
Record Dates: First submitted 2024-11-03; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia; Swallowing Disorder
Keywords: dysphagia; ultrasonography; swallowing assessment
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dysphagia patients: This cohort consists of patients with dysphagia undergoing swallowing function assessments. Participants will undergo two types of assessments: ultrasonography and fiberoptic endoscopic evaluation of swallowing (FEES), to evaluate key parameters of swallowing function.
  Interventions: Diagnostic Test: ultrasound evaluation; Diagnostic Test: Fiberoptic endoscopic evaluation of swallowing (FEES)

INTERVENTIONS:
Diagnostic Test: ultrasound evaluation — Use high-frequency ultrasonography to assess the swallowing function in patients with dysphagia. The ultrasound examination focuses on visualization of the pharyngeal region to measure vocal cord movement, swallowing reflex, pharyngeal contraction, and the presence and location of pharyngeal residue.
Diagnostic Test: Fiberoptic endoscopic evaluation of swallowing (FEES) — FEES involves the use of a flexible endoscope inserted through the nasal passage to observe the pharyngeal phase of swallowing directly. This procedure allows for the real-time assessment of key aspects of swallowing, including vocal cord function, swallowing reflex, pharyngeal contraction, and the detection of aspiration or penetration.

SUMMARY:
This study aims to explore the reliability of using ultrasonography (US) for the assessment of swallowing function in patients with dysphagia. The study will recruit 80 patients and compare the findings with those obtained from fiberoptic endoscopic evaluation of swallowing (FEES), which serves as the gold standard.

DETAILED DESCRIPTION:
This study will evaluate the reliability of using ultrasonography as a non-invasive tool for assessing swallowing function in patients with dysphagia. Participants will undergo US and FEES assessments to examine vocal cord function, swallowing reflex, pharyngeal contraction, aspiration/penetration, and stasis. The reliability, diagnostic accuracy, and inter-/intra-rater reliability will be analyzed to validate US as an effective alternative in clinical dysphagia assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older.
* Dysphagia patients referred for swallowing assessments.
* FOIS score between 2-6.

Exclusion Criteria:

* Unconscious patients or those unable to follow instructions.
* Unstable vital signs.
* Acute infections or mechanical ventilation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 years and older who have been referred for dysphagia evaluation. Participants will have varying degrees of swallowing difficulty, stemming from conditions such as stroke, head and neck cancer, or neurodegenerative diseases. Eligible individuals will have a Functional Oral Intake Scale (FOIS) score between 2 and 6. The population will be recruited from both outpatient and inpatient settings within the rehabilitation department of National Taiwan University Hospital. Patients must be conscious and able to follow instructions, ensuring accurate participation in both ultrasonography and fiberoptic endoscopic evaluation of swallowing (FEES). Those with unstable vital signs, acute infections, mechanical ventilation, or cognitive impairments preventing effective participation will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Reliability of Ultrasonography in Swallowing Function Assessment | Immediate post-assessment.
  Comparison with FEES findings

SECONDARY OUTCOMES:
Diagnostic Accuracy | Immediate post-assessment.
  Sensitivity, specificity, positive predictive value, and negative predictive value of US in detecting dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-mei Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsiao MY, Wu CH, Wang TG. Emerging Role of Ultrasound in Dysphagia Assessment and Intervention: A Narrative Review. Front Rehabil Sci. 2021 Aug 11;2:708102. doi: 10.3389/fresc.2021.708102. eCollection 2021. PMID 36188819
- [Background] Dunn CJ, Fitton A, Sorkin EM. Etidronic acid. A review of its pharmacological properties and therapeutic efficacy in resorptive bone disease. Drugs Aging. 1994 Dec;5(6):446-74. doi: 10.2165/00002512-199405060-00006. PMID 7858370
- [Background] Allen JE, Clunie GM, Winiker K. Ultrasound: an emerging modality for the dysphagia assessment toolkit? Curr Opin Otolaryngol Head Neck Surg. 2021 Jun 1;29(3):213-218. doi: 10.1097/MOO.0000000000000708. PMID 33741822